CLINICAL TRIAL: NCT01532648
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Budesonide MMX® 9 mg Extended-release Tablets as Add-on Therapy in Patients With Active, Mild or Moderate Ulcerative Colitis Not Adequately Controlled on a Background Oral 5-ASA Regimen
Brief Title: Randomized Placebo-Controlled Trial of Budesonide Multi-Matrix System (MMX®) 9 Milligrams (mg) in Participants With Ulcerative Colitis Currently on a 5-Aminosalicylic Acid (5-ASA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2011-0401
Record Dates: First submitted 2011-12-13; First posted 2012-02-14 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide MMX (Experimental): Participants will receive 1 oral tablet of budesonide MMX 9 mg for 56 days. Additionally, participants will continue to receive the same dose of their existing oral 5-ASA medication from their treating physician.
  Interventions: Drug: Budesonide MMX®; Drug: 5-ASA
- Placebo (Placebo Comparator): Participants will receive 1 oral tablet of matching budesonide MMX placebo for 56 days. Additionally, participants will continue to receive the same dose of their existing oral 5-ASA medication from their treating physician.
  Interventions: Drug: Placebo; Drug: 5-ASA

INTERVENTIONS:
Drug: Budesonide MMX® — Oral tablet taken daily in the morning after breakfast.
  Other Names: Budesonide Multi-Matrix System
  Arms: Budesonide MMX
Drug: Placebo — Matching budesonide MMX placebo oral tablet taken daily in the morning after breakfast.
  Arms: Placebo
Drug: 5-ASA — Acceptable oral 5-ASA medications to be received during the study include:
  * Asacol®, Asacol® HD, Lialda®, Pentasa® (generic: mesalamine), minimum daily dose ≥2.4 grams (g)
  * Azulfidine® (generic: sulfasalazine), minimum daily dose ≥4.0 g
  * Dipentum® (generic: olsalazine), minimum daily dose ≥2.0 g
  * Colazal®, Colazide® (generic: balsalazide), minimum daily dose ≥6.75 g

SUMMARY:
This study is to compare the efficacy and safety of budesonide MMX 9 mg versus placebo as add-on therapy to an existing oral 5-ASA regimen for the induction of remission in participants with active mild or moderate ulcerative colitis (UC).

DETAILED DESCRIPTION:
Eligible participants will be randomized to 1 of the following 2 treatment arms:

1. Budesonide MMX 9 mg (1 tablet)
2. Placebo (tablet indistinguishable from budesonide MMX 9 mg tablet)

The assigned study drug will be taken as a single oral tablet each morning after breakfast. In addition to the study drug, all participants will continue their existing background oral 5-ASA regimen during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years, inclusive.
2. Established diagnosis of UC, based on clinical history, exclusion of infectious causes, and characteristic endoscopic and histologic findings.
3. Active mild or moderate UC with an ulcerative colitis disease activity index (UCDAI) score ≥4 and ≤10, with a mucosal appearance score of ≥1, and physician's rating of disease activity of 1 or 2.
4. Experiencing active UC (flare) despite a therapeutic dose of an oral 5-ASA (for example, mesalamine ≥2.4 g/day for ≥6 weeks prior to randomization, or equivalent). At screening, photographic evidence of active UC based on mucosal appearance must be obtained.
5. Women of childbearing potential or men of reproductive potential must be willing to use an acceptable form of contraception.
6. Able to comprehend the full nature and purpose of the study, including possible risks and side effects, and also able to comply with all requirements of the study. Must be able to understand and voluntarily sign an informed consent prior to any study procedures.

Exclusion Criteria:

1. Limited distal proctitis (from anal verge to 15 centimeters [cm] above the pectineal line).
2. Severe UC (UCDAI >10 or physician global assessment [PGA] >2), or non-active UC (UCDAI <4).
3. Infectious colitis or any recent history of infectious colitis (within 30 days of Screening).
4. Active malignancy or carcinoma in situ within the last 5 years (treated non-melanoma skin cancers are not exclusionary).
5. Active ulcer or bleeding disorder that may affect evaluation of blood in the stool.
6. Evidence or history of toxic megacolon or bowel resection.
7. Crohn's disease or indeterminate colitis.
8. Known hypersensitivity to budesonide or any ingredients of the budesonide MMX tablets.
9. Active tuberculosis or other active systemic or local bacterial, fungal, or viral infection.
10. Liver cirrhosis, evident hepatic or renal disease or insufficiency, or significant impairment of the biohumoral parameters (≥2.5*upper limit of normal [ULN] for alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transpeptidase, or ≥2*ULN for creatinine). Elevations in bilirubin due to benign conditions such as Gilbert's syndrome are not exclusionary.
11. Severe diseases in other organs or systems.
12. Local or systemic complications or other pathological states requiring therapy with corticosteroids and/or immunosuppressive agents.
13. Type 1 diabetes.
14. Glaucoma or with a family history of glaucoma in first-degree relatives.
15. Known hepatitis B, hepatitis C, or human immunodeficiency virus (HIV), according to the local privacy policy.
16. Severe anemia (<9 g/deciliter [dL] hemoglobin), leukopenia (<2.5*10^9 white blood cells [WBC]/liter [L]), or granulocytopenia (<1.2*10^9 cells/L).
17. Participants with a history of pancolitis (disease that extends to the hepatic flexure or beyond) for ≥8 years or left-sided colitis (disease confined to the left colon [that is, distal to the splenic flexure]) ≥15 years who have not yet completed a surveillance colonoscopy for dysplasia/colorectal cancer screening within the past year.
18. Prior budesonide MMX treatment.
19. Use of oral corticosteroids including other budesonide formulations within the last 4 weeks prior to randomization.
20. Use of any rectal 5-ASA or corticosteroid formulations within the last 2 weeks prior to randomization.
21. Use of immunosuppressive agents within the last 8 weeks prior to randomization.
22. Use of anti-tumor necrosis factor-alpha (TNFα) agents or other biologic therapies within the last 3 months prior to randomization.
23. Participation in experimental therapeutic studies within 30 days of randomization (or within the last 3 months if in an anti-TNFα or biologic agent study). Note: participants who participated in observational-only studies (and who did not receive study therapy) are not excluded.
24. Any other medical condition that, in the Principal Investigator's opinion, would make the administration of the study drug or study procedures hazardous to the participant or obscure the interpretation of adverse events (AEs) by the appropriate independent ethics committee/institutional review board.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2012-01-27 (Actual); Primary Completion 2013-10-02 (Actual); Study Completion 2013-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Companies
Locations (114):
- United States (39):
  - Santarus Clinical Investigational Site 1043, Anaheim, California
  - Santarus Clinical Investigational Site 1071, Lakewood, California
  - Santarus Clinical Investigational Site 1003, San Diego, California
  - Santarus Clinical Investigational Site 1063, Littleton, Colorado
  - Santarus Clinical Investigational Site 1028, Bristol, Connecticut
  - Santarus Clinical Investigational Site 1035, Boynton Beach, Florida
  - Santarus Clinical Investigational Site 1045, Jacksonville, Florida
  - Santarus Clinical Investigational Site 1001, Largo, Florida
  - Santarus Clinical Investigational Site 1024, Maitland, Florida
  - Santarus Clinical Investigational Site 1029, Port Orange, Florida
  - Santarus Clinical Investigational Site 1010, Winter Park, Florida
  - Santarus Clinical Investigational Site 1002, Zephyrhills, Florida
  - Santarus Clinical Investigational Site 1050, Decatur, Georgia
  - Santarus Clinical Investigational Site 1075, Chicago, Illinois
  - Santarus Clinical Investigational Site 1065, Oak Lawn, Illinois
  - Santarus Clinical Investigational Site 1058, Indianapolis, Indiana
  - Santarus Clinical Investigational Site 1032, Shreveport, Louisiana
  - Santarus Clinical Investigational Site 1044, Annapolis, Maryland
  - Santarus Clinical Investigational Site 1016, Chesterfield, Michigan
  - Santarus Clinical Investigational Site 1081, Novi, Michigan
  - Santarus Clinical Investigational Site 1015, Wyoming, Michigan
  - Santarus Clinical Investigational Site 1068, Ypsilanti, Michigan
  - Santarus Clinical Investigational Site 1074, Rochester, Minnesota
  - Santarus Clinical Investigational Site 1061, Lebanon, New Hampshire
  - Santarus Clinical Investigational Site 1021, Cheektowaga, New York
  - Santarus Clinical Investigational Site 1072, Great Neck, New York
  - Santarus Clinical Investigational Site 1031, New York, New York
  - Santarus Clinical Investigational Site 1073, Wilmington, North Carolina
  - Santarus Clinical Investigational Site 1080, Cincinnati, Ohio
  - Santarus Clinical Investigational Site 1078, Cleveland, Ohio
  - Santarus Clinical Investigational Site 1082, Dayton, Ohio
  - Santarus Clinical Investigational Site 1064, Lancaster, Pennsylvania
  - Santarus Clinical Investigational Site 1006, Sayre, Pennsylvania
  - Santarus Clinical Investigational Site 1059, Austin, Texas
  - Santarus Clinical Investigational Site 1039, Houston, Texas
  - Santarus Clinical Investigational Site 1005, Pasadena, Texas
  - Santarus Clinical Investigational Site 1014, Lancaster, Utah
  - Santarus Clinical Investigational Site 1038, Chesapeake, Virginia
  - Santarus Clinical Investigational Site 1025, Christiansburg, Virginia
- Bulgaria (10):
  - Santarus Clinical Investigational Site 4003, Pleven
  - Santarus Clinical Investigational Site 4004, Plovdiv
  - Santarus Clinical Investigational Site 4009, Plovdiv
  - Santarus Clinical Investigational Site 4008, Rousse
  - Santarus Clinical Investigational Site 4001, Sofia
  - Santarus Clinical Investigational Site 4002, Sofia
  - Santarus Clinical Investigational Site 4005, Sofia
  - Santarus Clinical Investigational Site 4007, Sofia
  - Santarus Clinical Investigational Site 4010, Sofia
  - Santarus Clinical Investigational Site 4011, Sofia
- Canada (10):
  - Santarus Clinical Investigational Site 2003, Winnipeg, Manitoba
  - Santarus Clinical Investigational Site 2008, Halifax, Nova Scotia
  - Santarus Clinical Investigational Site 2004, London, Ontario
  - Santarus Clinical Investigational Site 2010, Ottawa, Ontario
  - Santarus Clinical Investigational Site 2002, Vaughan, Ontario
  - Santarus Clinical Investigational Site 2009, Montreal, Quebec
  - Santarus Clinical Investigational Site 2001, Sherbrooke, Quebec
  - Santarus Clinical Investigational Site 2007, Calgary
  - Santarus Clinical Investigational Site 2005, London
  - Santarus Clinical Investigational Site 2006, Québec
- Czechia (10):
  - Santarus Clinical Investigational Site 3001, Hradec Králové
  - Santarus Clinical Investigational Site 3006, Hradec Králové
  - Santarus Clinical Investigational Site 3005, Labem
  - Santarus Clinical Investigational Site 3003, Olomouc
  - Santarus Clinical Investigational Site 3004, Prague
  - Santarus Clinical Investigational Site 3007, Prague
  - Santarus Clinical Investigational Site 3009, Prague
  - Santarus Clinical Investigational Site 3002, Tábor
  - Santarus Clinical Investigational Site 3010, Ústí nad Orlicí
  - Santarus Clinical Investigational Site 3011, Valašské Meziříčí
- Santarus Clinical Investigational Site 8001, Tallinn, Estonia
- Hungary (11):
  - Santarus Clinical Investigational Site 5010, Békéscsaba
  - Santarus Clinical Investigational Site 5008, Budapest
  - Santarus Clinical Investigational Site 5009, Budapest
  - Santarus Clinical Investigational Site 5001, Debrecen
  - Santarus Clinical Investigational Site 5003, Gyula
  - Santarus Clinical Investigational Site 5004, Kaposvár
  - Santarus Clinical Investigational Site 5002, Miskolc
  - Santarus Clinical Investigational Site 5006, Mosonmagyaróvár
  - Santarus Clinical Investigational Site 5011, Pécs
  - Santarus Clinical Investigational Site 5005, Szeged
  - Santarus Clinical Investigational Site 5007, Vác
- Latvia (3):
  - Santarus Clinical Investigational Site 8101, Riga
  - Santarus Clinical Investigational Site 8102, Riga
  - Santarus Clinical Investigational Site 8103, Riga
- Lithuania (3):
  - Santarus Clinical Investigational Site 8202, Kaunas
  - Santarus Clinical Investigational Site 8201, Vilnius
  - Santarus Clinical Investigational Site 8203, Vilnius
- Poland (7):
  - Santarus Clinical Investigational Site 6003, Elblag
  - Santarus Clinical Investigational Site 6001, Krakow
  - Santarus Clinical Investigational Site 6002, Sopot
  - Santarus Clinical Investigational Site 6006, Szczecin
  - Santarus Clinical Investigational Site 6004, Warsaw
  - Santarus Clinical Investigational Site 6008, Warsaw
  - Santarus Clinical Investigational Site 6005, Warszawy
- Russia (13):
  - Santarus Clinical Investigational Site 9016, Lipetsk
  - Santarus Clinical Investigational Site 9005, Moscow
  - Santarus Clinical Investigational Site 9010, Moscow
  - Santarus Clinical Investigational Site 9004, Nizhny Novgorod
  - Santarus Clinical Investigational Site 9003, Ryazan
  - Santarus Clinical Investigational Site 9001, Saint Petersburg
  - Santarus Clinical Investigational Site 9008, Saint Petersburg
  - Santarus Clinical Investigational Site 9013, Saint Petersburg
  - Santarus Clinical Investigational Site 9014, Saint Petersburg
  - Santarus Clinical Investigational Site 9009, Saratov
  - Santarus Clinical Investigational Site 9007, Stavropol
  - Santarus Clinical Investigational Site 9006, Ufa
  - Santarus Clinical Investigational Site 9017, Volgograd
- Ukraine (7):
  - Santarus Clinical Investigational Site 7010, Crimea
  - Santarus Clinical Investigational Site 7002, Donetsk
  - Santarus Clinical Investigational Site 7001, Kharkiv
  - Santarus Clinical Investigational Site 7004, Kharkiv
  - Santarus Clinical Investigational Site 7006, Kyiv
  - Santarus Clinical Investigational Site 7008, Kyiv
  - Santarus Clinical Investigational Site 7005, Vinnytsia

REFERENCES:
- [Derived] Rubin DT, Cohen RD, Sandborn WJ, Lichtenstein GR, Axler J, Riddell RH, Zhu C, Barrett AC, Bortey E, Forbes WP. Budesonide Multimatrix Is Efficacious for Mesalamine-refractory, Mild to Moderate Ulcerative Colitis: A Randomised, Placebo-controlled Trial. J Crohns Colitis. 2017 Jul 1;11(7):785-791. doi: 10.1093/ecco-jcc/jjx032. PMID 28333362

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide MMX: Participants received 1 oral tablet of budesonide multi-matrix system (MMX) 9 milligrams (mg) for 56 days. Additionally, participants continued to receive the same dose of their existing oral 5-aminosalicylic acid (5-ASA) medication from their treating physician.
- Placebo: Participants received 1 oral tablet of matching budesonide MMX placebo for 56 days. Additionally, participants continued to receive the same dose of their existing oral 5-ASA medication from their treating physician.
Period: Overall Study
Arm/Group | Budesonide MMX | Placebo
Started | 255 | 255
Safety Population (All randomized participants who received at least 1 dose of study drug) | 255 | 255
Intent-To-Treat Population (Participants in Safety Population with active ulcerative colitis at study entry as cause of symptoms) | 230 | 228
Completed | 219 | 238
Not Completed | 36 | 17
Not completed — Lost to Follow-up | 3 | 4
Not completed — Lack of Efficacy | 4 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 12 | 9
Not completed — Withdrawal by Subject | 16 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug (Safety Population).
Groups:
- Budesonide MMX: Participants received 1 oral tablet of budesonide MMX 9 mg for 56 days. Additionally, participants continued to receive the same dose of their existing oral 5-ASA medication from their treating physician.
- Total: Total of all reporting groups
Arm/Group | Budesonide MMX | Placebo | Total
Number analyzed (Participants) | 255 | 255 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.86) | 44.9 (13.44) | 44.7 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 108 | 230
  Male | 133 | 147 | 280

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Clinical Remission at Day 56
Description: Clinical remission defined as a score of 0 for rectal bleeding and 0 for stool frequency components from the Ulcerative Colitis Disease Activity Index (UCDAI). UCDAI is the sum (0 to 12) of 4 severity scores (0 to 3). Stool frequency and rectal bleeding were based on information recorded in daily participant diaries. The diary entries were averaged for rectal bleeding and stool frequency for 3 days prior to (and closest to) Day 56 with non-missing diary data, within 5 days prior to (and closest to) Day 56. The 5 days did not include any days of the flexible sigmoidoscopy (or colonoscopy) or the preparation for the flexible sigmoidoscopy (or colonoscopy). These averages were rounded to integer values. If either subscore could not be calculated because of missing data, the score for that UCDAI component was set to missing. Participants with insufficient data at Day 56 were excluded from the analysis. Participants who had clinical remission at Baseline were classified as non-responders.
Time Frame: Baseline up to Day 56
Population: Participants who received at least 1 dose of study drug and had active ulcerative colitis (UC) at study entry as a cause of their symptoms (Intent-To-Treat Population [ITT]) with evaluable clinical remission data.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide MMX | Placebo
Number analyzed (Participants) | 230 | 228
Participants | 56 | 52

2. Secondary Outcome: Number of Participants of Who Achieved Clinical Response at Day 56
Description: Clinical response defined as an improvement in UCDAI from Baseline of ≥3 points with a rectal bleeding score ≤1. UCDAI is the sum (0 to 12) of 4 severity scores (0 to 3). Rectal bleeding was based on information recorded in daily participant diaries. The diary entries were averaged for rectal bleeding for 3 days prior to (and closest to) Day 56 with non-missing diary data, within 5 days prior to (and closest to) Day 56. The 5 days did not include any days of the flexible sigmoidoscopy (or colonoscopy) or the preparation for the flexible sigmoidoscopy (or colonoscopy). These averages were rounded to integer values. If either subscore could not be calculated because of missing data, the score for that UCDAI component was set to missing. Participants with insufficient data at Day 56 were excluded from the analysis.
Time Frame: Baseline up to Day 56
Population: Participants who received at least 1 dose of study drug and had active UC at study entry as a cause of their symptoms (ITT Population) with evaluable clinical response data.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide MMX | Placebo
Number analyzed (Participants) | 230 | 228
Participants | 101 | 86

3. Secondary Outcome: Number of Participants Who Achieved UCDAI Remission at Day 56
Description: UCDAI remission was defined as a total UCDAI score ≤1 with subscores of 0 for rectal bleeding, stool frequency, and mucosal appearance of the colon. UCDAI is the sum (0 to 12) of 4 severity scores (0 to 3). Stool frequency and rectal bleeding were based on information recorded in daily participant diaries and mucosal appearance was based on endoscopy results. The diary entries were averaged for rectal bleeding and stool frequency for 3 days prior to (and closest to) Day 56 with non-missing diary data, within 5 days prior to (and closest to) Day 56. The 5 days did not include any days of the flexible sigmoidoscopy (or colonoscopy) or the preparation for the flexible sigmoidoscopy (or colonoscopy). These averages were rounded to integer values. If the subscore could not be calculated because of missing data, the score for that UCDAI component was set to missing. Participants with insufficient data at Day 56 were excluded from the analysis.
Time Frame: Baseline up to Day 56
Population: Participants who received at least 1 dose of study drug and had active UC at study entry as a cause of their symptoms (ITT Population) with evaluable UCDAI remission data.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide MMX | Placebo
Number analyzed (Participants) | 230 | 228
Participants | 30 | 17

4. Secondary Outcome: Number of Participants Who Achieved Endoscopic Remission at Day 56
Description: Endoscopic remission was defined as a score of 0 in the mucosal appearance component subscore of the UCDAI at Day 56. UCDAI is the sum (0 to 12) of 4 severity scores (0 to 3). Mucosal appearance was based on endoscopy results. If the mucosal appearance subscore could not be calculated because of missing data, endoscopic remission was set to missing. Participants with insufficient data at Day 56 were excluded from the analysis.
Time Frame: Screening and Day 56
Population: Participants who received at least 1 dose of study drug and had active UC at study entry as a cause of their symptoms (ITT Population) with evaluable endoscopic response data.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide MMX | Placebo
Number analyzed (Participants) | 230 | 228
Participants | 46 | 28

5. Secondary Outcome: Number of Participants Who Achieved Histologic Healing at Day 56
Description: Participants achieved histologic healing if histologic assessments of all biopsy specimens were graded as 0 (normal mucosa). If the score for ≥1 sample was missing, the overall score at that visit was set to missing. Participants with insufficient data at Day 56 were excluded from analysis.
Time Frame: Baseline and Day 56
Population: Participants who received at least 1 dose of study drug and had active UC at study entry as a cause of their symptoms (ITT Population) with evaluable histologic healing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide MMX | Placebo
Number analyzed (Participants) | 230 | 228
Participants | 62 | 40

6. Secondary Outcome: Number of Participants With Treatment Failure at Day 56
Description: Treatment failure was defined as an unchanged, worsened, or missing UCDAI score at Day 56. UCDAI is the sum (0 to 12) of 4 severity scores (0 to 3). Stool frequency and rectal bleeding was based on information recorded in daily participant diaries and mucosal appearance was based on endoscopy results. The diary entries were averaged for rectal bleeding and stool frequency for 3 days prior to (and closest to) Day 56 with non-missing diary data, within 5 days prior to (and closest to) Day 56. The 5 days did not include any days of the flexible sigmoidoscopy (or colonoscopy) or the preparation for the flexible sigmoidoscopy (or colonoscopy). These averages were rounded to integer values. If the subscore could not be calculated because of missing data, the score for that UCDAI component was set to missing. Participants with insufficient data at Day 56 were excluded from the analysis.
Time Frame: Baseline up to Day 56
Population: Participants who received at least 1 dose of study drug and had active UC at study entry as a cause of their symptoms (ITT Population) with evaluable UCDAI data.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide MMX | Placebo
Number analyzed (Participants) | 230 | 228
Participants | 45 | 61

7. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease-Quality of Life (IBD-QoL) Questionnaire Scores
Description: The IBD-QoL questionnaire was self-completed by the participant. The IBD-QoL is a disease-specific instrument to evaluate the quality of life of participants with UC. This 32-item questionnaire has 4 dimensions: bowel function, emotional function, systemic symptoms, and social function. The total score is presented, which ranges from 32 to 224, with higher scores indicating a better quality of life. The scores of participants in remission usually range from 170 to 190. If >50% of the questionnaire answers for a particular dimension were missing, this dimension score was set to missing. The total score for the IBD-QoL was the sum of the domain scores, however, if any dimension score was missing, the total IBD-QoL score was set to missing.
Time Frame: Baseline, Days 14, 28, and 56
Population: Participants who received at least 1 dose of study drug and had active UC at study entry as a cause of their symptoms (ITT Population) with evaluable IBD-QoL data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Budesonide MMX | Placebo
Number analyzed (Participants) | 230 | 228
scores on a scale
  Baseline: number analyzed (Participants) | 230 | 226
  Baseline | 132.8 (31.36) | 134.1 (32.48)
  Change at Day 14: number analyzed (Participants) | 228 | 224
  Change at Day 14 | 24.4 (27.45) | 21.3 (29.20)
  Change at Day 28: number analyzed (Participants) | 230 | 225
  Change at Day 28 | 31.8 (33.38) | 25.7 (33.16)
  Change at Day 56: number analyzed (Participants) | 230 | 225
  Change at Day 56 | 31.1 (38.73) | 31.7 (37.02)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 85
Description: All randomized participants who received at least 1 dose of study drug (Safety Population).
Arm/Group | Budesonide MMX | Placebo
Serious Adverse Events (participants affected / at risk) | 10/255 | 2/255
Other Adverse Events (participants affected / at risk) | 14/255 | 14/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide MMX (N=255) | Placebo (N=255)
Colitis ulcerative (Gastrointestinal disorders) | 6 | 1
Pancreatitis active (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide MMX (N=255) | Placebo (N=255)
Colitis ulcerative (Gastrointestinal disorders) | 11 | 9
Acne (Skin and subcutaneous tissue disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.